CLINICAL TRIAL: NCT04724135
Title: Assessment of Menopause Related Quality of Life Among Health Professionals in University Hospitals of UMC in Nur-Sultan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nazarbayev University Medical Center (Other)
Collaborators: University of South Florida (Other); Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Gauri Bapayeva, Principal Investigator, Nazarbayev University Medical Center
Organization: Nazarbayev University (Other)
Other Study IDs: 024-2020
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Menopause
Keywords: Menopause; Quality of life; Healthcare providers
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Female health-care givers aged 45 to 64 years. The study participants will be recruited from UMC (Clinical Academic Department (CAD) of Women's Health, Pediatric Clinical Academic Department, Republic Diagnostic Center (RDC) and National Center for Children's Rehabilitation (NCCR)), Nur-Sultan, Kazakhstan.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The first part will assess the sociodemographic variables and reproductive characteristics, and the second part contain the Menopause-Specific Quality of Life (MENQOL) questionnaire The 29 questions of the MENQOL are divided into four domains: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29).

SUMMARY:
This study aims to investigate the quality of life of menopausal health-care providers in University Medical Center (UMC) hospitals in Nur-Sultan and identify whether there is a difference in the quality of life between two major groups of women health-care professionals: physicians and nurses, and to explore factors influencing on it.

DETAILED DESCRIPTION:
Quality of life has turned into a reference for the so-called "state of wellbeing" that includes six domains: physical health, social relationships, psychological state, spiritual concerns, environmental features, and level of independence. Quality of life is perceived as a major health component, especially for menopausal women, and has become an essential research topic that has been discussed widely in the literature.

Therefore, from the HRQoL perspective, the consequences of the climacterium should be considered as a specific aspect of health-related quality of life in studies that include this segment of the population. The increased life expectancy of the general population and of women in particular, has turned women's health care in this phase of life into a priority; the way this should be accomplished, however, represents one of the main sources of public health debate.

Quality of work life is a comprehensive and general schema, which is essential in improving specialized personnel's satisfaction and attracting and preserving personnel. It also results in positive theories such as increasing profits and provocation. Nevertheless, although physicians and nurses are expected to provide patient care and improve their quality of life, their own needs and their own quality of life have been either largely underestimated or ignored.

Providing care in these cases is very demanding in physical, emotional, and spiritual terms. Their work requires certain qualities, such as empathy, compassion, and closeness to the individuals and families they care for. Therefore, daily work may be significantly influenced by the menopausal transition, especially in nurses and physicians Work is beneficial for menopausal women by providing fulfilment, self-esteem, identity and social needs. But working environments like those with lack of temperature control, cramped conditions, some uniforms and stress can also make menopause symptoms worse. Menopause refers to the time when a woman's menstrual period stops for 12 consecutive months after the last period and is characterized by a decline in the production of the ovarian hormones, mainly estrogen and progesterone. The lack of these hormones makes some women prone to experiencing common symptoms that include, but are not limited to, sleep disorders, mood alterations, hot flashes, depression, urinary tract infections, vaginal infections, and increased risk for osteoporosis and cardiovascular diseases. Providing up-to-date information to women about menopause, its management, and the use of menopausal hormone therapy (MHT) may serve as an important step towards treating postmenopausal symptoms thereby improving the QOL of postmenopausal women.

According to a recent study, the level of awareness and knowledge of women about the menopause is directly proportional to their ability to control their symptoms as menopausal symptoms can have a negative impact on work but menopause in the workplace still remains a taboo. This study aims to investigate the QoL of menopausal health-care providers in UMC hospitals in Nur-Sultan and identify whether there is a difference in the quality of life between two major groups of women health-care professionals: physicians and nurses, and to explore factors influencing on it.

ELIGIBILITY:
Inclusion Criteria:

* We will include all menopausal health-care providers working in CAD of Women's Health and Pediatric CAD UMC, NCCR, and RDC, Nur-Sultan Kazakhstan. In order to get the highest possible response rate as well as evaluate the non-response bias, there is a need to follow-up to those who did not responded.

Exclusion Criteria:

* Women with serious health problems, such as severe chronic diseases, including psychological/psychiatric comorbidities, and use of specific drugs for them, will not be included in the study

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Since this study is aimed to investigate and determine the quality of life in menopausal women, the participants are menopausal women aged 45 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Menopause Quality of Life Measurement | 36 month
  The participants will be asked to indicate whether they had experienced symptoms or problems within the past month and, if so, to rate how bothersome they were on a seven-point Likert scale from 0 to 6: with 0 indicating that they were not at all bothered and 6 indicating that they were extremely bothered. The 29 questions of the MENQOL (supported by NCBI and NHI) are divided into four domains: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29).

CONTACTS AND LOCATIONS:
Overall Officials: Milan Terzic, MD, PhD, Study Director — Nazarbayev University Medical Center; Sanja Terzic, MD, Study Director — Nazarbayev University Medical Center; Gauri Bapayeva, MD, PhD, Principal Investigator — Nazarbayev University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided